CLINICAL TRIAL: NCT06250049
Title: Effectiveness of the Implementation of a Standardized Foot Care Protocol in Individuals With Diabetes in Primary Care in Salamanca
Brief Title: Improvement of Diabetic Foot Care in Salamanca Through the Implementation of Standardized Protocols.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Marta Manzano Garcia, Principal investigator, Sanidad de Castilla y León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GRS/2534/B/22
Record Dates: First submitted 2024-01-12; First posted 2024-02-08 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Primary Health Care; Diabetes; Diabetic Foot
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group of patients will be attended according to a diabetic foot care protocol implemented in Primary Care in Salamanca. In addition, those patients and/or caregivers will receive group education sessions on Diabetic Foot Care at the Health Centers.
  Interventions: Other: Diabetic foot care protocol; Other: Group education sessions for patients and/or caregivers
- Control Group (No Intervention): Usual care

INTERVENTIONS:
Other: Diabetic foot care protocol — Introduction of the diabetic foot care protocol in Primary Care in Salamanca, sensitization, and training of nursing professionals in Health Centers (HC).
  Arms: Intervention Group
Other: Group education sessions for patients and/or caregivers — Conducting group education sessions for patients and/or caregivers on Diabetic Foot Care at the Health Centers.
  Arms: Intervention Group

SUMMARY:
Introduction: Diabetic foot (DF) is among the most prevalent complications affecting individuals with diabetes. In Salamanca, 25,631 individuals are enrolled in the Diabetes Care Service, with only 3.06% undergoing a foot examination.

Objective: To evaluate the effectiveness of implementing a standardized foot care protocol for individuals with diabetes, accompanied by a sensitization and training strategy for nursing professionals.

Methodology: Quasi-experimental pre- and post-study with a control group conducted in the Health Centers of Salamanca.

Population: Patients included in the Diabetes Care Service (306) (12,458 men and 11,348 women).

Measurements:

In professionals: number of professionals involved and satisfaction level. In diabetic individuals: Sociodemographic, anthropometric, lifestyle, and clinical variables related to disease control will be measured, along with variables related to protocol implementation (percentage of diabetics who have undergone foot examination, Ankle-Brachial Index (ABI), risk stratification and foot monitoring, percentage of individuals with DF, percentage of individuals with healed DF ulcers, and percentage of individuals who have undergone amputation). Improvement in quality of life will be measured using the COOP-WONCA questionnaire.

Expected outcomes: It is anticipated that this study will provide evidence regarding the relationship between protocol implementation and an increase in the detection and care of at-risk feet and DF, as well as an improvement in the quality of life of individuals with diabetes.

DETAILED DESCRIPTION:
The diabetic foot (DF) is a common complication in individuals with DM, significantly increasing morbidity and mortality. Patients with DM face a 10-20 times higher relative risk of lower limb amputation than those without diabetes, primarily due to ulcers or previous injuries associated with neuropathy and peripheral arterial disease, termed DF (WHO, 2020). Short-to-medium-term mortality post-amputation is comparable to, or even higher than, many cancers (Armstrong et al., 2020).

Diabetic foot disease (DFD) causes significant patient suffering and imposes a substantial burden on caregivers, healthcare professionals, health services, and society at large (Schaper et al., 2020). Despite its impact, DFD is often underestimated and underdiagnosed, as healthcare professionals perceive its prevalence and clinical, social, and economic consequences inadequately (Suárez and Lozano, 2014). In Spain, DF screening and risk stratification are systematically conducted in Primary Care (PC), but overall data show a low percentage of DF examinations and record-keeping in medical records, with significant variations among autonomous communities, potentially influenced by the implementation of strategies addressing this complication (Ministry of Health, 2022).

To address existing barriers hindering more equitable and high-quality care for DF patients within the National Health System (NHS), the document "Diabetic Foot Management" is developed as part of the Diabetes Strategy (Ministry of Health, 2022). Based on the International Working Group on the Diabetic Foot (IWGDF) consensus, it incorporates key recommendations from various guidelines regarding educational aspects (for patients, caregivers, and professionals), DF screening, and interventions to reduce amputations and enhance the quality of life. It emphasizes that DF management should primarily occur in Primary Care, adopting a multidisciplinary approach (Ministry of Health, 2022).

ELIGIBILITY:
Inclusion Criteria:

* Individuals included in the "Care for individuals with DM" Service of the Primary Care Services Portfolio of SACYL, aged 14 years and older.

Exclusion Criteria:

* Change of patient's residence to another Health Area.
* Patient who voluntarily declines to be included.
* Patients with amputation of both lower limbs.
* Patient's decease.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25631 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of individuals with diabetes mellitus who have undergone examination and exploration of both feet | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes mellitus who have undergone examination and exploration of both feet.
Number of individuals with diabetes who have undergone foot risk stratification. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes who have undergone foot risk stratification.
Number of individuals with diabetes who have received group education related to diabetic foot care. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes who have received group education related to diabetic foot care.
Quality of life of individuals with diabetes | Pre (baseline period) and Post-intervention (6-month)
  Quality of life of individuals with diabetes pre and post intervention measured through the COOP-WONCA questionnaire. The COOP/WONCA questionnaire was originally developed by a group of primary care physicians at The Darmouth Primary Care Cooperative Information Project (COOP Project), Hanover, New Hampsshire USA. The questionnaire consists of 9 items with a 5-point Likert-type scale. , where higher scores express worse levels of functioning. It was in 1988 when the World Organization of National Colleges, Academies, and Academic Associations of General Practitioners/Family Physicians (WONCA) adopted this instrument.
Number of individuals with diabetes with a nursing care plan established. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes with a nursing care plan established.
Number of individuals with diabetes who have received individual education related to diabetic foot care. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes who have received individual education related to diabetic foot care.

SECONDARY OUTCOMES:
Number of Primary Care teams where the sensitization and training strategy has been implemented. | Post-intervention (6-month)
  Number of Primary Care teams where the sensitization and training strategy has been implemented.
Satisfaction level of professionals regarding sensitization and training | Post-intervention (6-month)
  Satisfaction level of professionals regarding sensitization and training through an ad hoc questionnaire carried out by the Ministry of Health of the Government of Castilla y León (SACYL) with a Likert-type scale.
Percentage of professionals who have implemented the protocol after training. | Pre (baseline period) and Post-intervention (6-month)
  Percentage of professionals who have implemented the protocol after training.
Number of individuals detected with at-risk feet. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals detected with at-risk feet.
Number of individuals detected with diabetic foot. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals detected with diabetic foot.
Number of individuals with diabetes with diabetic foot ulcers who have achieved healing (at least one) in the last year. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes with diabetic foot ulcers who have achieved healing (at least one) in the last year.
Number of individuals with diabetes who have undergone lower limb amputation (partial or total) in the last year. | Pre (baseline period) and Post-intervention (6-month)
  Number of individuals with diabetes who have undergone lower limb amputation (partial or total) in the last year.
Number of diabetic individuals referred to podiatry, vascular surgery, and traumatology and orthopedics. | Pre (baseline period) and Post-intervention (6-month)
  Number of diabetic individuals referred to podiatry, vascular surgery, and traumatology and orthopedics.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Manzano García, Principal Investigator — Sanidad de Castilla y León
Locations (1):
- Marta Manzano García, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No